CLINICAL TRIAL: NCT06008080
Title: VISTA Nova Study (Navitor Post-Market Clinical Follow Up Study)
Brief Title: Post-Market Clinical Follow Up Study With Navitor Valve
Acronym: VISTA Nova
Status: Recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10476
Record Dates: First submitted 2023-08-16; First posted 2023-08-23 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Aortic Stenosis
Keywords: NAVITOR; Transcatheter aortic valve implantation (TAVI); Aortic Stenosis; Cardiovascular Disease
MeSH Terms: conditions — Aortic Valve Stenosis; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Navitor Transcatheter Aortic Valve, FlexNav Delivery System, Navitor Loading System: The Navitor valve is available in five valve sizes to cover annulus diameters from 19 mm to 30 mm. The FlexNav delivery system is available in two sizes, small and large. The Navitor loading system is an accessory used to compress and load the Navitor valve onto the FlexNav delivery system and is available in two sizes, small and LG+.
  Interventions: Device: Navitor Transcatheter Aortic Valve, FlexNav Delivery System, Navitor Loading System

INTERVENTIONS:
Device: Navitor Transcatheter Aortic Valve, FlexNav Delivery System, Navitor Loading System — Subjects will undergo transcatheter aortic valve replacement (TAVR) with the Navitor valve, the FlexNav Delivery system and the Navitor Loading System

SUMMARY:
Evaluation of the safety and performance of the Navitor TAVI System in a Global Study

DETAILED DESCRIPTION:
The VISTA Nova Study will evaluate the safety, performance, and long-term durability of the Navitor valve in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Patient is eligible per the current approved indication after Heart Team discussion and intended to undergo a Navitor TAVI procedure.
* The patient has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent as approved by the IRB (Investigational Review Board)/EC (Ethics Committee) of the respective clinical site.
* The patient and the treating physician agree that the subject will return for all required post procedure follow up visits.

Exclusion Criteria:

* Patient is not eligible for the Navitor TAVI System per the current Instructions for Use (IFU)
* Life expectancy < 12 months from the time of informed consent due to non-cardiac co-morbid conditions.
* In the judgment of the Investigator, patient presents with a medical, social, or psychological condition that could limit the ability or willingness to participate in the study, comply with study required testing and/or follow-up visits or that could impact scientific integrity of the study.
* Known contraindication for computed tomography (CT) or sensitivity to contrast media, which cannot be adequately premedicated.
* Inability to tolerate antiplatelet/anticoagulation therapy or nitinol alloy (nickel and titanium), which cannot be adequately premedicated.
* Currently participating in an investigational drug or device study that may confound the results of this study
* Anatomy that makes insertion and endovascular access to the aortic valve difficult and/or impossible

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll subjects of all genders from the population of patients qualifying for TAVI.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality at 30 days post-TAVI procedure | 30 days post index procedure
  Death from all causes at 30 days post-TAVI procedure
Moderate or greater paravalvular leak at 30 days post-TAVI procedure | 30 days post index procedure
  Assessment of paravalvular leak at 30 days post-TAVI procedure

CONTACTS AND LOCATIONS:
Overall Officials: Alper Öner, MD, Principal Investigator — Universitätsmedizin Rostock, Germany; Nicolas Dumonteil, MD, Principal Investigator — Clinique Pasteur Toulouse, France
Locations (35):
- Royal Hobart Hospital, Hobart, Australia
- France (4):
  - Clinique du Millénaire, Montpellier
  - Mutualiste Montsouris, Paris
  - CHRU Hopital de Pontchaillou, Rennes
  - Clinique Pasteur Toulouse, Toulouse
- Germany (10):
  - Herz- u. Gefäßzentrum Bad Bevensen, Bad Bevensen
  - Deutsches Herzzentrum der Charité, Berlin
  - St Johannes Hospital Dortmund, Dortmund
  - Kliniken der Friedrich-Alexander-Universitat, Erlangen
  - Klinikum der Johann Wolfgang Goethe-Universität Frankfurt, Frankfurt
  - UKE Hamburg, Hamburg
  - Universitätsklinikum Schleswig-Holstein - Campus Kiel, Kiel
  - Deutsches Herzzentrum München des Freistaates Bayern, München
  - University Hospital Rostock, Rostock
  - Universitätsklinikum Ulm, Ulm
- Italy (5):
  - Az. Osp. Spedali Civili di Brescia, Brescia
  - Casa di Cura Pineta Grande, Castel Volturno
  - Centro Cardiologico Monzino, Milan
  - Ospedale San Raffaele - Cardiac, Milan
  - Policlinico San Donato, San Donato Milanese
- Onze Lieve Vrouw Gasthuis, Amsterdam, Netherlands
- ULS de Lisboa Ocidental, Carnaxide, Portugal
- Spain (7):
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Hospital General Juan Ramon Jimenez, Huelva
  - Hospital de Gran Canaria Doctor Negrín, Las Palmas
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Consorcio Hospital General Universitario de Valencia, Valencia
- Sahlgrenska University Hospital - Gothenburg, Gothenburg, Sweden
- KS St. Gallen / USZ, Sankt Gallen, Switzerland
- United Kingdom (4):
  - Kings College Hospital, London
  - James Cook University Hospital, Middlesbrough
  - Royal Stoke University Hospital, Stoke-on-Trent
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: No